CLINICAL TRIAL: NCT02138981
Title: Hepatic Resection Versus Transarterial Chemoembolization as the Initial Treatment for Resectable Hepatocellular Carcinoma Beyond Milan Criteria
Brief Title: Hepatectomy Versus Chemoembolization for Resectable Hepatocellular Carcinoma Beyond Milan Criteria
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Kaiping Central Hospital (Other); First People's Hospital of Chenzhou (Other); Dongguan Shi People's Hospital (Unknown)
Responsible Party: Principal Investigator, Shi Ming, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCC_S012
Record Dates: First submitted 2014-05-13; First posted 2014-05-15 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Resectable Hepatocellular Carcinoma Beyond Milan Criteria
Keywords: Hepatocellular Carcinoma; Milan Criteria
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate Resection (Active Comparator): patients received immediate surgical hepatic resection
  Interventions: Procedure: Immediate Resection
- Chemoembolization and Response-Dependent Resection (Experimental): patients underwent transarterial chemoembolization (TACE) as initial treatments, and only patients who showed good response were subjected to surgical resection.
  Interventions: Procedure: Chemoembolization and Response-Dependent Resection

INTERVENTIONS:
Procedure: Chemoembolization and Response-Dependent Resection — patients underwent transarterial chemoembolization (TACE) as initial treatments, and only patients who showed good response were subjected to surgical resection.
  Arms: Chemoembolization and Response-Dependent Resection
Procedure: Immediate Resection — patients received immediate surgical resection.
  Arms: Immediate Resection

SUMMARY:
The purpose of this study is to compare the survival outcomes between hepatic resection and transarterial lipiodol chemoembolization (TACE) used as the initial treatment in patients with Resectable Hepatocellular Carcinoma Beyond Milan Criteria.

DETAILED DESCRIPTION:
For patients with large/multiple, and resectable hepatocellular carcinomas (HCCs) without macrovascular invasion or extrahepatic spread, the choice of treatment remains largely controversial. For these patients, transarterial lipiodol chemoembolization (TACE) is recommended as a palliative therapy.

On the other hand, many authors still believe that hepatic resection is the only potential curative treatment in these patients because it is still feasible to remove all macroscopic tumors safely at surgery. With advances in surgical techniques, more large/multiple HCCs are now resectable, and long-term results have been reported that ranged from 30% to 58% at 5 years; even patients with large bilobar multiple HCC could reach a survival rate of more than 20% at 5 years after hepatic resection.

Until now, there have been only a few studies that compared the outcomes of hepatic resection and TACE in the treatment of multiple HCCs, and these have reported controversial results. Some studies showed that hepatic resection had survival benefi t over TACE, but other studies showed the opposite result ( 11-15 ). Therefore, the investigators performed this prospective study in consecutive patients with large/multiple, and resectable HCCs to compare the outcomes in patients who underwent hepatic resection or TACE as the initial treatment.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of HCC based on the diagnostic criteria for HCC used by the European Association for the Study of the Liver (EASL).
* The patient has not been previously treated with surgery, radiation therapy, radiofrequency ablation, percutaneous ethanol or acetic acid injection, or cryoablation.
* The tumor beyound milan criteria.
* The tumor was evaluated to be resectable by a same group of surgeon.
* Patients must have at least one tumor lesion that can be accurately measured according to EASL criteria
* No serious concurrent medical illness
* Not pregnant or breast-feeding patients
* Cirrhotic status of Child-Pugh class A only
* The following laboratory parameters:

  * Platelet count ≥ 80,000/µL
  * Hemoglobin ≥ 8.5 g/dL
  * Total bilirubin ≤ 1.5 mg/dL Serum albumin ≥ 35 g/L
  * ASL and AST ≤ 5 x upper limit of normal
  * Serum creatinine ≤ 1.5 x upper limit of normal
  * INR ≤ 1.5 or PT/APTT within normal limits
  * Absolute neutrophil count (ANC) >1,500/mm3
* Ability to understand the protocol and to agree to and sign a written informed consent document

Exclusion Criteria:

* Tumor vascular invasion or distant metastases
* Significant renal impairment (creatinine clearance < 30 mL/minute) or patients on dialysis
* On anticoagulation or suffering from a known bleeding disorder
* Unstable coronary artery disease or recent MI
* Known history of HIV
* History of organ allograft
* Known or suspected allergy to the investigational agents or any agent given in association with this trial.
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry.
* Any other hemorrhage/bleeding event > CTCAE Grade 3 within 4 weeks of first dose of study drug
* Serious non-healing wound, ulcer, or bone fracture
* Known central nervous system tumors including metastatic brain disease
* severe Arterioportal Shunts or Arteriavein Shunts

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 436 (Estimated)
Dates: Start 2014-05-01; Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
overall survival time | 5 years

SECONDARY OUTCOMES:
disease free survival | 5 years
Number of Adverse Events | 30 days
  All severe adverse events for the entire course of treatment, including treatment for primary tumor and recurrent tumor.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Shi, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Cancer Center Sun Yat-sen University, Guangzhou, Guangdong, China